CLINICAL TRIAL: NCT03254498
Title: Is Endocuff Vision Assisted Colonoscopy Superior to Cap Assisted Colonoscopy to Detect Adenomas
Brief Title: Detection in Tandem Endocuff Cap Trial
Acronym: DETECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RD15/061
Record Dates: First submitted 2017-08-14; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Colonic Neoplasms; Adenomas Serrated; Colo-rectal Cancer; Colon Adenoma
Keywords: colonic adenoma; serrated polyps; caecal intubation time; withdrawal time; polyp miss rate
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: It is a randomised back to back study to compare the performance of cap assisted colonoscopy (CAC) and Endocuff assisted colonoscopy (EAC)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endocuff assisted colonoscopy (Active Comparator): Participants are randomised to undergo first either with Endocuff or cap assisted colonoscopy during colonoscopy.
  Interventions: Device: Endocuff
- Cap assisted colonoscopy (Placebo Comparator): Participants are randomised to undergo first either with Endocuff or cap assisted colonoscopy during colonoscopy.
  Interventions: Device: cap assisted colonoscopy (CAC)

INTERVENTIONS:
Device: Endocuff — It is a randomised back to back study to compare cap and Endocuff to detect adenoma in colonoscopic examination
  Arms: Endocuff assisted colonoscopy
Device: cap assisted colonoscopy (CAC) — cap assisted colonoscopy (CAC)
  Arms: Cap assisted colonoscopy

SUMMARY:
A randomised back to back study comparing cap and Endocuff to detect adenomas during colonoscopy

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and over
2. Referral for surveillance, or diagnostic colonoscopy
3. Ability to give informed consent

Exclusion Criteria:

1. Absolute contraindications to colonoscopy
2. Established or suspicion of large bowel obstruction or pseudo-obstruction
3. Known colon cancer or polyposis syndromes
4. Known colonic strictures
5. Known severe diverticular segment (that is likely to impede colonoscope passage)
6. Patients with active colitis (ulcerative colitis, Crohn's colitis, diverticulitis, infective colitis)
7. Patients lacking capacity to give informed consent
8. Pregnancy
9. Patients who are on clopidogrel, warfarin, or other new generation anticoagulants who have not stopped this for the procedure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Adenoma miss rate | 1 day
  Comparison of adenoma miss rate between cap ( CAC) and Endocuff assisted colonoscopy(E

SECONDARY OUTCOMES:
Mean adenoma per procedure | 1 day
  Difference in mean adenomas detected per procedure (MAP) between EAC and CAC.
Endocuff or cap exchange | 1 day
  Number of times Cap or Endocuff are removed to complete the procedure
Ceacal intubation and withdrawal time | 1 day
  Comparison of caecal intubation and withdrawal time
miss rate of advanced polyps | 1 day
  Comparison of miss rates of advanced adenomas, serrated polyps and proxima polyps between CAC and EAC
Comfort score | 1 day
  Comparison of patient comfort score between CAC and EAC

OTHER OUTCOMES:
comparison of surveillance intervals | Once histology is available usually takes 10-14 days
  To compare any surveillance interval difference between CAC and EAC

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Saunders, MD, Principal Investigator — St Mark's Hospital, Northwest London Hospitals NHS Trust
Locations (1):
- NorthWest London Hospitals - NOrthwick park hospital, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rameshshanker R, Tsiamoulos Z, Wilson A, Rajendran A, Bassett P, Tekkis P, Saunders BP. Endoscopic cuff-assisted colonoscopy versus cap-assisted colonoscopy in adenoma detection: randomized tandem study-DEtection in Tandem Endocuff Cap Trial (DETECT). Gastrointest Endosc. 2020 Apr;91(4):894-904.e1. doi: 10.1016/j.gie.2019.11.046. Epub 2019 Dec 10. PMID 31836474